CLINICAL TRIAL: NCT03882047
Title: Efficacy and Safety of Mometasone Furoate Aqueous Nasal Spray vs Placebo and Flonase® (Fluticasone Propionate) in Seasonal Allergic Rhinitis Patients (I94-001)
Brief Title: Mometasone Furoate Aqueous (MK-0887/SCH 032088) Nasal Spray vs Placebo and FLONASE® in Seasonal Allergic Rhinitis Patients (I94-001)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: I94-001; I94-001 (Other: Schering-Plough Protocol Number)
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Results first posted 2019-09-06 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Rhinitis, Allergic, Seasonal
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Mometasone Furoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Both participant and investigator were blinded to treatment identity. Because the mometasone furoate and fluticasone propionate bottles were not identical in appearance, a double-dummy study design was used and each bottle had a matching placebo. Thus, although participants received bottles of different appearance, they did not know whether bottles contained active substance or placebo.
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mometasone furoate nasal spray (Experimental): Participants receive 200 mcg of mometasone furoate nasal spray and fluticasone propionate placebo matching nasal spray once daily.
  Interventions: Drug: Mometasone furoate; Drug: Fluticasone propionate placebo
- Fluticasone propionate nasal spray (Active Comparator): Participants receive 200 mcg of fluticasone propionate nasal spray and mometasone furoate placebo matching nasal spray once daily.
  Interventions: Drug: Fluticasone propionate; Drug: Mometasone furoate placebo
- Placebo nasal spray (Placebo Comparator): Participants receive mometasone furoate placebo matching nasal spray and fluticasone propionate placebo matching nasal spray once daily.
  Interventions: Drug: Mometasone furoate placebo; Drug: Fluticasone propionate placebo

INTERVENTIONS:
Drug: Mometasone furoate — Mometasone furoate nasal spray, 200 mg once daily
  Other Names: NASONEX®; MK-0887; SCH 032088
  Arms: Mometasone furoate nasal spray
Drug: Fluticasone propionate — Fluticasone propionate nasal spray, 200 mg once daily
  Other Names: FLONASE®
  Arms: Fluticasone propionate nasal spray
Drug: Mometasone furoate placebo — Mometasone furoate placebo matching nasal spray, once daily
  Arms: Fluticasone propionate nasal spray; Placebo nasal spray
Drug: Fluticasone propionate placebo — Fluticasone propionate placebo matching nasal spray, once daily
  Arms: Mometasone furoate nasal spray; Placebo nasal spray

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of mometasone furoate (SCH 32088) aqueous nasal spray 200 mcg once daily compared to placebo once daily in the treatment of participants with seasonal allergic rhinitis. Flonase (fluticasone propionate) nasal spray 200 mcg once daily has been chosen as the active control for this study.

ELIGIBILITY:
Inclusion Criteria:

* 2-year history of seasonal allergic rhinitis
* Positive skin test response to a local seasonal allergen (current, or performed in investigator's office within the past year)
* Good health and free of any unstable, clinically significant disease, other than allergic rhinitis, that would interfere with the study schedule or evaluation of seasonal allergic rhinitis

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Women of childbearing potential who are not using an acceptable form of birth control
* Significant history of metabolic, cardiovascular, neurologic, hematologic, hepatic, gastrointestinal, cerebrovascular, respiratory, or renal disease, or any other disorder which, in the judgment of the investigator, could interfere with the study, or require treatment which might interfere with the study
* Use of any chronic medication which could affect the course of seasonal allergic rhinitis
* Asthma requiring chronic use of inhaled or systemic corticosteroids (inhaled bronchodilators are permitted for asthma treatment)
* Current or history of frequent, clinically significant sinusitis or chronic purulent postnasal drip
* Upper respiratory tract or sinus infection that requires antibiotic therapy within the previous 2 weeks, or a viral upper respiratory infection (URI) within the 7 days prior to Screening
* Dependence upon nasal, oral or ocular decongestants, or nasal topical antihistamines, in the opinion of the investigator
* Has rhinitis medicamentosa
* Investigational drug use within the previous 30 days
* Nasal structural abnormalities, including large nasal polyps and marked septal deviation, that significantly interfere with nasal air flow
* Immunotherapy (desensitization therapy), unless on a stable maintenance schedule for at least one month prior to the Screening visit
* History of multiple drug allergies, allergy to antihistamines or corticoids
* History of psychosis, antagonistic personality, poor motivation, hypochondriasis, or any other emotional or intellectual problems that are likely to limit the validity of consent to participate in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 1994-08-11 (Actual); Primary Completion 1994-09-16 (Actual); Study Completion 1994-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Groups:
- Mometasone Furoate Nasal Spray: Participants received 200 mcg of mometasone furoate nasal spray and fluticasone propionate placebo matching nasal spray once daily for 14 days.
- Fluticasone Propionate Nasal Spray: Participants received 200 mcg of fluticasone propionate nasal spray and mometasone furoate placebo matching nasal spray once daily for 14 days.
- Placebo Nasal Spray: Participants receive mometasone furoate placebo matching nasal spray and fluticasone propionate placebo matching nasal spray once daily for 14 days.
Period: Overall Study
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Started | 104 | 105 | 104
Treated | 104 | 104 | 103
Completed | 98 | 95 | 88
Not Completed | 6 | 10 | 16
Not completed — Adverse Event | 0 | 2 | 2
Not completed — Treatment Failure | 3 | 3 | 12
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Did Not Wish to Continue | 1 | 4 | 1
Not completed — Noncompliance With Protocol | 2 | 0 | 0
Not completed — Did Not Meet Eligibility | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 104 | 104 | 103 | 311
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.72 (10.61) | 30.88 (10.71) | 31.14 (11.62) | 31.25 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 53 | 39 | 141
  Male | 55 | 51 | 64 | 170

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Nasal Symptom Score Averaged Over Day 1 Through Day 15 (Based on Participant Diaries)
Description: Change from baseline averaged over study Day 1 through study Day 15 was calculated for Total Nasal Symptom Score, based on participant diaries. Participants scored 4 symptoms (rhinorrhea, stuffiness, itching, sneezing) in their diaries using the following scale: 0=none, 1=mild, 2=moderate, 3=severe. The Total Nasal Symptom Score was the sum of the 4 individual scores (range=0-12; higher score indicating more frequent/severe nasal symptoms.) Change from baseline was the 15-day average score minus the baseline score. Scores were recorded twice daily, in the morning (AM) and night (PM). Average AM/PM scores were first calculated separately, then averaged together to obtain the 15-day average score. Baseline score was an average of the 3 AM scores and 3 PM scores preceding treatment. Negative changes indicated a decrease in symptom severity.
Time Frame: Baseline and Day 1 through Day 15 (averaged over 15 days)
Population: All randomized participants who completed at least one valid post-baseline visit and had available diary data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 104 | 104 | 103
Score on a scale | -2.8 (2.2) | -3.4 (2.3) | -0.9 (2.3)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.03, ANOVA

2. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score at Day 4 (Physician Evaluation)
Description: Change from baseline at Day 4 was calculated for the Total Nasal Symptom Score, as assessed by the physician. The Total Nasal Symptom Score was a composite of the following symptoms: rhinorrhea, nasal stuffiness, nasal itching, and sneezing scores. The physician scored each symptom during the study visit on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. The composite score ranged from 0-12. Change from baseline = visit score - baseline score (Day 1 visit). A negative change from baseline score indicated a decrease in symptom severity.
Time Frame: Baseline (Day 1) and Day 4
Population: All randomized participants who completed at least one valid post-baseline visit and had available Day 4 visit data for Total Nasal Symptom Score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 103 | 104 | 103
Score on a scale | -3.2 (2.8) | -3.5 (3.0) | -1.8 (2.9)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.31, ANOVA

3. Secondary Outcome: Change From Baseline in the Total Nasal Symptom Score at Day 15 (Physician Evaluation)
Description: Change from baseline at Day 15 was calculated for the Total Nasal Symptom Score, as assessed by the physician. The Total Nasal Symptom Score was a composite of the following symptoms: rhinorrhea, nasal stuffiness, nasal itching, and sneezing scores. The physician scored each symptom during the study visit on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. The composite score ranged from 0-12. Change from baseline = visit score - baseline score (Day 1 visit). A negative change from baseline score indicated a decrease in symptom severity.
Time Frame: Baseline (Day 1) and Day 15
Population: All randomized participants who completed at least one valid post-baseline visit and had available Day 15 visit data for Total Nasal Symptom Score.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 95 | 95 | 88
Score on a scale | -4.4 (2.9) | -5.5 (2.7) | -2.7 (3.3)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.01, ANOVA

4. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis at Day 4 (Physician Evaluation)
Description: Change from baseline at Day 4 was calculated for the Overall Condition of Seasonal Allergic Rhinitis, as assessed by the physician. The physician scored their overall condition on study Day 4 on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity of symptoms. Change from baseline = visit score - baseline score (Day 1 visit). A negative change from baseline score indicated a decrease in symptom severity.
Time Frame: Baseline (Day 1) and Day 4
Population: All randomized participants who completed at least one valid post-baseline visit and had available Day 4 data for Overall Condition of Seasonal Allergic Rhinitis (physician evaluated).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 103 | 104 | 103
Score on a scale | -0.5 (0.7) | -0.7 (0.8) | -0.3 (0.7)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = 0.08, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.10, ANOVA

5. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis at Day 15 (Physician Evaluation)
Description: Change from baseline at Day 15 was calculated for the overall condition of seasonal allergic rhinitis, as assessed by the physician. The physician scored their overall condition on study Day 15 on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity of symptoms. Change from baseline = visit score - baseline score (Day 1 visit). A negative change from baseline score indicated a decrease in symptom severity.
Time Frame: Baseline (Day 1) and Day 15
Population: All randomized participants who completed at least one valid post-baseline visit and had available Day 15 data for Overall Condition of Seasonal Allergic Rhinitis (physician evaluated)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 95 | 95 | 88
Score on a scale | -0.9 (0.8) | -1.2 (0.8) | -0.5 (0.9)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.01, ANOVA

6. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis at Day 4 (Participant Evaluation)
Description: The overall condition of seasonal allergic rhinitis was evaluated by the participant on Day 4, based on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity of symptoms. Change from baseline = visit score - baseline score (Day 1 visit). A negative change from baseline score indicated a decrease in symptom severity.
Time Frame: Baseline (Day 1) and Day 4
Population: All randomized participants who completed at least one valid post-baseline visit and had available Day 4 data for Overall Condition of Seasonal Allergic Rhinitis (participant evaluation).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 103 | 104 | 103
Score on a scale | -0.6 (0.8) | -0.8 (0.7) | -0.3 (0.8)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p = 0.02, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.05, ANOVA

7. Secondary Outcome: Change From Baseline in Overall Condition of Seasonal Allergic Rhinitis at Day 15 (Participant Evaluation)
Description: The overall condition of seasonal allergic rhinitis was evaluated by the participant on Day 15, based on the following scale: 0=none, 1=mild, 2=moderate; and 3=severe. A higher value indicated greater severity of symptoms. Change from baseline = visit score - baseline score (Day 1 visit). A negative change from baseline score indicated a decrease in symptom severity.
Time Frame: Baseline (Day 1) and Day 15
Population: All randomized participants who completed at least one valid post-baseline visit and had available Day 15 data for Overall Condition of Seasonal Allergic Rhinitis (participant evaluation)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 95 | 95 | 88
Score on a scale | -1.1 (0.8) | -1.3 (0.8) | -0.5 (0.9)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.06, ANOVA

8. Secondary Outcome: Response to Therapy at Day 4 (Physician Evaluation)
Description: Response to therapy was assessed by evaluating the participant's relief of nasal symptoms at Day 4. The physician evaluated the participant's response using the following 5-point scale: 1=complete relief, 2=marked relief, 3=moderate relief, 4=slight relief, and 5=no relief. The scores were averaged across each treatment group, with a lower score indicating a greater response to therapy and an improvement in nasal symptoms.
Time Frame: Day 4
Population: All randomized participants who completed at least one valid post-baseline visit and had available Day 4 data for Response to Therapy (physician evaluation).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 103 | 104 | 103
Score on a scale | 3.2 (0.9) | 3.1 (1.1) | 3.8 (1.0)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.46, ANOVA

9. Secondary Outcome: Response to Therapy at Day 15 (Physician Evaluation)
Description: Response to therapy was assessed by evaluating the participant's relief of nasal symptoms at Day 15. The physician evaluated the participant's response using the following 5-point scale: 1=complete relief, 2=marked relief, 3=moderate relief, 4=slight relief, and 5=no relief. The scores were averaged across each treatment group, with a lower score indicating a greater response to therapy and an improvement in nasal symptoms.
Time Frame: Day 15
Population: All randomized participants who completed at least one valid post-baseline visit and had available Day 15 data for Response to Therapy (physician evaluation).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 95 | 95 | 88
Score on a scale | 2.7 (1.1) | 2.4 (1.1) | 3.2 (1.3)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.07, ANOVA

10. Secondary Outcome: Response to Therapy at Day 4 (Participant Evaluation)
Description: Response to therapy was evaluated by participants and based upon their status scored at Day 4. Participants evaluated their response to therapy using the following 5-point scale: 1 = Complete Relief, 2 = Marked Relief, 3 = Moderate Relief, 4= Slight Relief, and 5 = Treatment Failure. The scores were averaged across each treatment group, with a lower score indicating a greater response to therapy and an improvement in nasal symptoms.
Time Frame: Day 4
Population: All randomized participants who completed at least one valid post-baseline visit and had available Day 4 data for Response to Therapy (participant evaluation).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 103 | 104 | 103
Score on a scale | 3.2 (0.9) | 3.1 (1.1) | 3.7 (1.1)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.53, ANOVA

11. Secondary Outcome: Response to Therapy at Day 15 (Participant Evaluation)
Description: Response to therapy was evaluated by participants and based upon their status scored at Day 15. Participants evaluated their response to therapy using the following 5-point scale: 1 = Complete Relief, 2 = Marked Relief, 3 = Moderate Relief, 4= Slight Relief, and 5 = Treatment Failure. The scores were averaged across each treatment group, with a lower score indicating a greater response to therapy and an improvement in nasal symptoms.
Time Frame: Day 15
Population: All randomized participants who completed at least one valid post-baseline visit and had available Day 15 data for Response to Therapy (participant evaluation).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 95 | 95 | 88
Score on a scale | 2.6 (1.1) | 2.4 (1.1) | 3.4 (1.3)
Statistical Analysis 1: Comparison: Mometasone Furoate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 2: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Test type: Other; p < 0.01, ANOVA
Statistical Analysis 3: Comparison: Mometasone Furoate Nasal Spray vs Fluticasone Propionate Nasal Spray; Test type: Other; p = 0.12, ANOVA

ADVERSE EVENTS:
Time Frame: Up to 45 days
Description: All randomized participants who received at least one dose of study treatment and had at least one post-baseline evaluation for safety.
Arm/Group | Mometasone Furoate Nasal Spray | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/104 | 0/103
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/104 | 0/103
Other Adverse Events (participants affected / at risk) | 30/104 | 24/104 | 28/103
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mometasone Furoate Nasal Spray (N=104) | Fluticasone Propionate Nasal Spray (N=104) | Placebo Nasal Spray (N=103)
FATIGUE (General disorders) | 1 (1) | 4 (5) | 6 (13)
HEADACHE (Nervous system disorders) | 14 (19) | 13 (23) | 18 (28)
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 (12) | 7 (9) | 4 (6)
NASAL DISCOMFORT (Respiratory, thoracic and mediastinal disorders) | 7 (14) | 6 (16) | 4 (8)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 2 (3) | 4 (7)

LIMITATIONS AND CAVEATS:
AE Preferred Terms were converted from WHO-ART dictionary to the MedDRA version 12.0.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has 30 days prior to submission for publication or presentation to review copies of abstracts or manuscripts for publication (including texts of oral presentations) which report any results of the Protocol study. Sponsor shall have editorial rights with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation with regard to proprietary information and the accuracy of the information contained in the publication.